CLINICAL TRIAL: NCT03779503
Title: A Clinical Comparison of Two Daily Disposable Soft Contact Lenses
Brief Title: Comparison of Two Daily Disposable Soft Contact Lenses
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: CooperVision, Inc. (Industry)
Responsible Party: Sponsor
Organization: CooperVision International Limited (CVIL) (Industry)
Allocation: Randomized | Model: Crossover | Masking: Double | Purpose: Treatment
Other Study IDs: EX-MKTG-99 (C18-649)
Record Dates: First submitted 2018-12-13; First posted 2018-12-19 (Actual); Results first posted 2020-10-08 (Actual); Last update posted 2020-10-08 (Actual); Status verified 2020-09

CONDITIONS: Astigmatism Bilateral

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: Yes | US Export: Yes

ARMS (2):
- midafilcon A (Active Comparator): Subjects will be randomized to wear midafilcon A 1 day for one week of daily wear during the study.
  Interventions: Device: midafilcon A
- somofilcon A (Active Comparator): Subjects will be randomized to wear somofilcon A 1 day for one week of daily wear during the study.
  Interventions: Device: somofilcon A

INTERVENTIONS:
Device: midafilcon A — midafilcon A 1 day daily disposable contact lens
  Arms: midafilcon A
Device: somofilcon A — somofilcon A 1 day daily disposable contact lens
  Arms: somofilcon A

SUMMARY:
The aim of this study was to investigate the short-term clinical performance and subjective acceptance of the two study lenses.

DETAILED DESCRIPTION:
This study was a randomised, double-masked, crossover, bilateral dispensing study, controlled by cross-comparison. Fifty-five subjects will wear each lens brand for approximately one week in random order. Lenses were worn on a daily wear, daily disposable basis.

ELIGIBILITY:
Inclusion Criteria:

1. They are between 18 and 40 years of age (inclusive).
2. They understand their rights as a research subject and are willing to sign a Statement of Informed Consent.
3. They are willing and able to follow the protocol.
4. They are an existing silicone hydrogel reusable spherical contact lens wearer in both eyes.
5. They have a contact lens spherical prescription between -0.25D and -6.00D (inclusive) based on ocular refraction.
6. They own a wearable pair of spectacles and wear them on the day of the initial visit.
7. At dispensing, they can attain at least 0.20 logMAR distance high contrast visual acuity in each eye with the study lenses within the available power range.
8. They are willing to comply with the wear schedule (at least five days per week and for at least eight hours per day).
9. They agree not to participate in other clinical research for the duration of the study.

Exclusion Criteria:

1. They have an ocular disorder, which would normally contra-indicate contact lens wear.
2. They have a systemic disorder, which would normally contra-indicate contact lens wear.
3. They are using any topical medication such as eye drops or ointment, or use any rewetting/lubricating drops whilst on this study.
4. They are aphakic.
5. They have had corneal refractive surgery.
6. They have any corneal distortion resulting from previous hard or rigid lens wear or have keratoconus.
7. They are pregnant or breastfeeding.
8. They have any ocular abnormality which would, in the opinion of the investigator, normally contraindicate contact lens wear
9. They have any infectious disease which would, in the opinion of the investigator, contraindicate contact lens wear or pose a risk to study personnel; or they have any immunosuppressive disease (e.g. HIV), or a history of anaphylaxis or severe allergic reaction.
10. They have taken part in any contact lens or care system clinical research within two weeks prior to starting this study.

Ages: 18 Years to 40 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 55 (Actual)
Dates: Start 2019-02-08 (Actual); Primary Completion 2019-07-30 (Actual); Study Completion 2019-09-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Philip Morgan, PhD MCOptom FAAO FBCLA, Principal Investigator — Eurolens Research
Locations (1):
- CooperVision Inc., Pleasanton, California, United States

RESULTS

PARTICIPANT FLOW:
Groups:
- Midafilcon A Then Somofilcon A: Subjects will be randomized to wear midafilcon A 1 day for one week of daily wear the cross-over to somofilcon A for one week of daily wear during the study.
  midafilcon A: midafilcon A 1 day daily disposable contact lens somofilcon A: somofilcon A 1 day daily disposable contact lens
- Somofilcon A Then Midafilcon A: Subjects will be randomized to wear somofilcon A 1 day for one week of daily wear then cross-over to midafilcon A for one week of daily wear during the study.
  somofilcon A: somofilcon A 1 day daily disposable contact lens midafilcon A: midafilcon A 1 day daily disposable contact lens
Period: First Intervention
Arm/Group | Midafilcon A Then Somofilcon A | Somofilcon A Then Midafilcon A
Started | 28 | 27
Completed | 27 | 26
Not Completed | 1 | 1
Not completed — Adverse Event | 0 | 1
Not completed — Withdrawal by Subject | 1 | 0
Period: Second Intervention
Arm/Group | Midafilcon A Then Somofilcon A | Somofilcon A Then Midafilcon A
Started | 27 | 26
Completed | 27 | 26
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Groups:
- Overall Study: Subjects were randomized to wear either midafilcon A 1 day or somofilcon A 1 day for one week of daily wear the cross-over to the other for one week of daily wear during the study.
  midafilcon A: midafilcon A 1 day daily disposable contact lens somofilcon A: somofilcon A 1 day daily disposable contact lens
Arm/Group | Overall Study
Number analyzed (Participants) | 55
Age, Categorical [Count of Participants; unit: Participants]
  <=18 years | 0
  Between 18 and 65 years | 55
  >=65 years | 0
Age, Continuous [Mean (Standard Deviation); unit: years] | 26.3 (6.3)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 47
  Male | 8
Race and Ethnicity Not Collected [Count of Participants; unit: Participants] — Population: Race and Ethnicity were not collected from any participant.
Region of Enrollment [Number; unit: participants]
  United States | 55

OUTCOME MEASURES:

1. Primary Outcome: Lens Fit - Horizontal Centration
Description: Assessment of horizontal centration of lens (extremely nasal, slightly nasal, optimum, slightly temporal, extremely temporal)
Time Frame: Baseline
Measure: Number; unit: percentage of lenses
Arm/Group | Midafilcon A | Somofilcon A
Number analyzed (Participants) | 54 | 54
percentage of lenses
  Extremely nasal | 0 | 0
  Slightly nasal | 6 | 4
  Optimum | 61 | 48
  Slightly Temporal | 33 | 48
  Extremely Temporal | 0 | 0

2. Primary Outcome: Lens Fit - Horizontal Centration
Description: as for outcome 1
Time Frame: One Week
Measure: Number; unit: participants of lenses
Arm/Group | Midafilcon A | Somofilcon A
Number analyzed (Participants) | 53 | 53
participants of lenses
  Extremely nasal | 0 | 0
  Slightly nasal | 8 | 6
  Optimum | 60 | 55
  Slightly Temporal | 32 | 40
  Extremely Temporal | 0 | 0

3. Primary Outcome: Lens Fit - Vertical Centration
Description: Assessment of vertical centration of lens (extremely inferior, slightly inferior, optimum, slightly superior, extremely superior)
Time Frame: Baseline
Measure: Number; unit: percentage of lenses
Arm/Group | Midafilcon A | Somofilcon A
Number analyzed (Participants) | 54 | 54
percentage of lenses
  Extremely inferior | 0 | 0
  Slightly inferior | 31 | 22
  Optimum | 54 | 46
  Slightly Superior | 15 | 31
  Extremely Superior | 0 | 0

4. Primary Outcome: Lens Fit - Vertical Centration
Description: as for outcome 3
Time Frame: One Week
Measure: Number; unit: percentage of lenses
Arm/Group | Midafilcon A | Somofilcon A
Number analyzed (Participants) | 53 | 53
percentage of lenses
  Extremely inferior | 2 | 0
  Slightly inferior | 32 | 26
  Optimum | 47 | 43
  Slightly Superior | 19 | 30
  Extremely Superior | 0 | 0

5. Primary Outcome: Lens Fit - Corneal Coverage
Description: Assessment of corneal coverage of lens (extremely inadequate, slightly inadequate, optimum, slightly excessive, extremely excessive)
Time Frame: Baseline
Measure: Number; unit: percentage of lenses
Arm/Group | Midafilcon A | Somofilcon A
Number analyzed (Participants) | 54 | 54
percentage of lenses
  Extremely inadequate | 0 | 0
  Slightly inadequate | 17 | 22
  Optimum | 76 | 70
  Slightly excessive | 7 | 7
  Extremely excessive | 0 | 0

6. Primary Outcome: Lens Fit - Corneal Coverage
Description: as for outcome 5
Time Frame: One Week
Measure: Number; unit: percentage of lenses
Arm/Group | Midafilcon A | Somofilcon A
Number analyzed (Participants) | 53 | 53
percentage of lenses
  Extremely inadequate | 2 | 0
  Slightly inadequate | 19 | 34
  Optimum | 72 | 60
  Slightly excessive | 8 | 6
  Extremely excessive | 0 | 0

7. Primary Outcome: Lens Fit - Lens Movement
Description: Lens movement assessed per corneal coverage (extremely inadequate, slightly inadequate, optimum, slightly excessive, extremely excessive)
Time Frame: Baseline
Measure: Number; unit: percentage of lenses
Arm/Group | Midafilcon A | Somofilcon A
Number analyzed (Participants) | 54 | 54
percentage of lenses
  Extremely inadequate | 0 | 0
  Slightly inadequate | 11 | 9
  Optimum | 56 | 79
  Slightly excessive | 33 | 13
  Extremely excessive | 0 | 0

8. Primary Outcome: Lens Fit - Lens Movement
Description: as for outcome 7
Time Frame: One Week
Measure: Number; unit: percentage of lenses
Arm/Group | Midafilcon A | Somofilcon A
Number analyzed (Participants) | 53 | 53
percentage of lenses
  Extremely inadequate | 0 | 0
  Slightly inadequate | 13 | 11
  Optimum | 55 | 75
  Slightly excessive | 30 | 13
  Extremely excessive | 2 | 0

9. Secondary Outcome: Subjective Score for Vision
Description: Subjects will score on visual analogue scale for vision (0 -100) (0 - Unacceptable, 20 - Very poor, 40 - Poor, 60 - Good, 80 - Very Good, 100 - Excellent)
Time Frame: Baseline
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Midafilcon A | Somofilcon A
Number analyzed (Participants) | 54 | 54
units on a scale | 93.1 (8.5) | 95.0 (8.6)

10. Secondary Outcome: Subjective Score for Vision
Description: as for outcome 9
Time Frame: One week
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Midafilcon A | Somofilcon A
Number analyzed (Participants) | 53 | 53
units on a scale | 86.5 (15.5) | 91.7 (12.2)

ADVERSE EVENTS:
Time Frame: From dispense up to one week for each study lenses, a total of two weeks
Arm/Group | Midafilcon A | Somofilcon A
All-Cause Mortality (participants affected / at risk) | 0/55 | 0/55
Serious Adverse Events (participants affected / at risk) | 0/55 | 0/55
Other Adverse Events (participants affected / at risk) | 0/55 | 0/55

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2018-09-25): https://cdn.clinicaltrials.gov/large-docs/03/NCT03779503/Prot_SAP_001.pdf